CLINICAL TRIAL: NCT05576415
Title: An Open-Label, Multiple-Dose Clinical Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of OC-01 (Varenicline Solution) Nasal Spray in Adult Chinese Subjects With Dry Eye Disease
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of OC-01 in Adult Chinese With Dry Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX03003
Record Dates: First submitted 2022-09-27; First posted 2022-10-12 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye Disease
Keywords: OC-01 (Varenicline Solution); Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Nasal Sprays

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OC-01 (Experimental)
  Interventions: Drug: Varenicline Tartrate Nasal Spray

INTERVENTIONS:
Drug: Varenicline Tartrate Nasal Spray — Intranasal delivery of OC-01 (varenicline solution) 0.6 mg/mL twice a day (BID) for 28 days.
  Other Names: OC-01 (varenicline solution) Nasal Spray

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics (PK) in adult Chinese subjects with dry eye disease (DED)1 after bilateral nasal spray administration of OC-01 (varenicline solution) Nasal Spray at a concentration of 0.6 mg/mL.

ELIGIBILITY:
Inclusion Criteria:

Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to the Screening Visit

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery) or extraocular surgery in either eye within three months or refractive surgery (e.g., laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within 12 months of the Screening Visit
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, acute conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or investigational product components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Cmax of varenicline after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively. | Visit 1 [Day 1]: From predose of the 1st dosing to 12 hours post-dose. Visit 3 [Day 28]: From predose of the last dosing to 120 hours post-dose.
  To evaluate the Cmax of varenicline in adult Chinese with dry eye disease (DED) after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively.
Tmax of varenicline after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively. | Visit 1 [Day 1]: From predose of the 1st dosing to 12 hours post-dose. Visit 3 [Day 28]: From predose of the last dosing to 120 hours post-dose.
  To evaluate the Tmax of varenicline in adult Chinese subjects with DED after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively.
AUCtau(Area under the concentration-time curve during a dosing interval) of varenicline after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively. | Visit 1 [Day 1]: From predose of the 1st dosing to 12 hours post-dose. Visit 3 [Day 28]: From predose of the last dosing to 120 hours post-dose.
  To evaluate the AUCtau of varenicline in adult Chinese subjects with DED after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively.
AUC0-last(Area under the concentration-time curve from time 0 to the time of the last measured non-zero concentration) of varenicline after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively. | Visit 1 [Day 1]: From predose of the 1st dosing to 12 hours post-dose. Visit 3 [Day 28]: From predose of the last dosing to 120 hours post-dose.
  To evaluate the AUC0-last of varenicline in adult Chinese subjects with DED after the first dosing at Visit 1 [Day 1] and after the last dosing at Visit 3 [Day 28], respectively.
T1/2 of varenicline after the last dosing at Visit 3 [Day 28] | Visit 3 [Day 28]: From predose of the last dosing to 120 hours post-dose
  To evaluate the T1/2 of varenicline after the last dosing at Visit 3 [Day 28] in adult Chinese subjects with DED.
λz of varenicline after the last dosing at Visit 3 [Day 28] | Visit 3 [Day 28]: From predose of the last dosing to 120 hours post-dose
  To evaluate the λz of varenicline after the last dosing at Visit 3 [Day 28] in adult Chinese subjects with DED.

SECONDARY OUTCOMES:
Change from baseline in Schirmer's Test Score (STS) at Visit 1 [Day 1], Visit 2 [Day 14] and Visit 3 [Day 28] | From Day 1 to Day 28
  To assess the Schirmer's Test Score (STS) using Schirmer's strips in adult Chinese subjects with DED after bilateral nasal spray administration of OC-01 (varenicline solution) Nasal Spray at a concentration of 0.6 mg/mL.
  For STS, the minimum value is 0.0mm, the maximum value is 35.0mm, the higher scores of change mean a better outcome.
Change from baseline in Eye Dryness Score (EDS) at Visit 2 [Day 14] and Visit 3 [Day 28] | From Day 14 to Day 28
  To assess the Eye Dryness Score (EDS) using a Visual Analog Scale (VAS) in adult Chinese subjects with DED after bilateral nasal spray administration of OC-01 (varenicline solution) Nasal Spray at a concentration of 0.6 mg/mL.
  For EDS, the minimum value is 0mm, the maximum value is 100mm, the higher scores of change mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: LU, Doctor, Principal Investigator — Huashan Hospital; ZHANG, Doctor, Principal Investigator — Huashan Hospital; DING, Study Director — Corxel Pharmaceuticals
Locations (1):
- Huashan Hospital, Shanghai, China